CLINICAL TRIAL: NCT05795959
Title: Ensuring Precision-Medicine Delivery for Veterans With Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 67785
Record Dates: First submitted 2023-03-09; First posted 2023-04-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
Keywords: Precision Medicine; Lung Diseases; Lay health worker; Veteran health
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to this arm of the study will receive usual care with supplemental education and support provided by a lay VA volunteer trained on evidence-based lung cancer care.
  Interventions: Behavioral: Receive education on precision medicine
- Control (No Intervention): Participants randomized to this arm of the study will receive usual clinical care.

INTERVENTIONS:
Behavioral: Receive education on precision medicine — Patients who consent to participating in the study and are randomized to the intervention group, will meet 1 on 1 with a trained lay VA volunteer. The trained lay VA volunteer will conduct phone calls with patients until the end of the 1 month enrollment period to deliver education regarding precision medicine.
  Arms: Intervention

SUMMARY:
The goal of this study is to learn if using a lay VA volunteer, who will assist patients with education regarding precision medicine, can improve care quality and outcomes for Veteran patients with lung cancer.

DETAILED DESCRIPTION:
Participants in the intervention group will receive 1:1 communication with a lay VA volunteer in addition to their usual clinical care. The lay VA volunteer will provide patients with education about precision medicine and support in their care. Researchers will compare a control group who will receive their usual oncology care as provided by clinical teams at the VA. There will be no change in their care.

All participants will be asked to complete a survey at the time of enrollment in the study, and also at 1 month. This survey will measure patient participation in their cancer care, satisfaction with healthcare decisions, and overall questions about knowledge of precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years old that have been newly diagnosed with any stage of lung cancer.
* Patients must have the ability to understand and willingness to provide verbal consent.
* Participants must speak English.

Exclusion Criteria:

* Inability to consent to the study, severe mental illness (e.g. schizophrenia) or institutionalization.
* Patients who anticipate moving care outside the Veterans Affairs Palo Alto Health Care System within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Knowledge of precision medicine for cancer care from time of enrollment to 1 month post-enrollment | Baseline
  Using 8 multiple choice items adapted from an 8-item survey tool, Knowledge and Purpose of Molecular Profiling, by Davies et. al., 2020, we will assess knowledge of precision medicine for cancer care at time of enrollment and again at 1-month post-enrollment. For example one question asks 'tumor testing is helpful for guiding the treatment of lung cancer,' with answer choices: yes or no. Answers will be scored as number or percent correct.

SECONDARY OUTCOMES:
Patient activation using the "Patient Activation Measure" survey | Baseline
  Each patient will receive a validated patient activation survey using the "Patient Activation Measure" at baseline. This is a validated measure from Insignia Health. Responses are: disagree strongly, disagree, agree, agree strongly with higher activation correlated with responses of agree and agree strongly. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-10, minimum score is 0 (if all not-applicable) and maximum is 100. Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining "Behaviors and Pushing Further. Scores for each group will be averaged at baseline.
Patient activation using the "Patient Activation Measure" survey | 1 month post-enrollment
  Each patient will receive a validated patient activation survey using the "Patient Activation Measure" at 1 month post-enrollment. This is a validated measure from Insignia Health. Responses are: disagree strongly, disagree, agree, agree strongly with higher activation correlated with responses of agree and agree strongly. Each item is rated on 4-point scale (1 strongly disagree to 4 strongly agree, with additional "not applicable" option). Higher scores indicate greater patient activation. For the PAM-10, minimum score is 0 (if all not-applicable) and maximum is 100. Raw scores are converted into activation levels per the scoring guidelines by Insignia Health for: level 1 Disengaged and Overwhelmed, level 2 Becoming Aware but Still Struggling, level 3 Taking Action and Gaining Control, level 4 Maintaining "Behaviors and Pushing Further. Scores for each group will be averaged at 1 month post-enrollment
Patient Satisfaction With Shared Decision Making using the "Shared Decision Making Questionnaire" Survey | Baseline
  Using 9 items of the validated 9-item Shared Decision Making Questionnaire (SDM-Q-9) at baseline. Responses are "completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, or completely agree," with 1=completely disagree and 6= completely agree. Higher scores indicate greater levels of satisfaction.
Patient Satisfaction With Shared Decision Making using the "Shared Decision Making Questionnaire" Survey | 1 month post-enrollment
  Using 9 items of the validated 9-item Shared Decision Making Questionnaire (SDM-Q-9) at 1 month post-enrollment. Responses are "completely disagree, strongly disagree, somewhat disagree, somewhat agree, strongly agree, or completely agree," with 1=completely disagree and 6= completely agree. Higher scores indicate greater levels of satisfaction.
Receipt of molecular testing | 6 months post-enrollment
  Chart review will be used to abstract whether participants received molecular testing
Receipt of targeted therapy for those with an eligible molecular target | 6 months post-enrollment
  Chart review will be used to abstract whether participants with a molecular target received targeted treatment for the molecular target

CONTACTS AND LOCATIONS:
Overall Officials: Manali I Patel, MD MPH MS, Principal Investigator — VA Palo Alto
Locations (1):
- VA Palo Alto, Palo Alto, California, United States